CLINICAL TRIAL: NCT04318236
Title: Multifactorial Randomised Trial Investigating Outcome and Adherence Relevant Factors in an Online Problem-solving Self-help Intervention for Mild and Moderate Depressive Symptoms
Brief Title: Factorial Trial Investigating Outcome and Adherence Relevant Factors in an Online Self-help Intervention for Depression
Acronym: HERMES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: KEK BE 2019-01795
Record Dates: First submitted 2020-03-17; First posted 2020-03-23 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Depression Mild; Depression Moderate
MeSH Terms: interventions — RBPMS protein, human; Counseling

STUDY DESIGN:
Intervention Model Description: Multifactorial design (factorial trial), following the Multiphase optimisation Strategy (MOST)
Who Masked: Participant
Masking Description: Participants only know that the delivery or the context of online interventions are to be improved and investigated. However, they don't know the exact interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Online-Program + factors 1,2,3,4 (Experimental): In this "arm" all four factors are set to "active" (i.e. yes):
  * diagnostic interview
  * motivational module
  * guidance
  * e-mail reminders
  Interventions: Behavioral: HERMES (Online Self-Help Intervention based on problem-solving therapy)
- Online-Program + factors 1,2,3 (Experimental): In this "arm" three factors are set to "active" (i.e. yes):
  * diagnostic interview
  * motivational module
  * guidance
  Interventions: Behavioral: HERMES (Online Self-Help Intervention based on problem-solving therapy)
- Online-Program + factors 1,2,4 (Experimental): In this "arm" three factors are set to "active" (i.e. yes):
  * diagnostic interview
  * motivational module
  * e-mail reminders
  Interventions: Behavioral: HERMES (Online Self-Help Intervention based on problem-solving therapy)
- Online-Program + factors 1,2 (Experimental): In this "arm" two factors are set to "active" (i.e. yes):
  * diagnostic interview
  * motivational module
  Interventions: Behavioral: HERMES (Online Self-Help Intervention based on problem-solving therapy)
- Online-Program + factors 1,3,4 (Experimental): In this "arm" three factors are set to "active" (i.e. yes):
  * diagnostic interview
  * guidance
  * e-mail reminders
  Interventions: Behavioral: HERMES (Online Self-Help Intervention based on problem-solving therapy)
- Online-Program + factors 1,3 (Experimental): In this "arm" two factors are set to "active" (i.e. yes):
  * diagnostic interview
  * guidance
  Interventions: Behavioral: HERMES (Online Self-Help Intervention based on problem-solving therapy)
- Online-Program + factors 1,4 (Experimental): In this "arm" two factors are set to "active" (i.e. yes):
  * diagnostic interview
  * e-mail reminders
  Interventions: Behavioral: HERMES (Online Self-Help Intervention based on problem-solving therapy)
- Online-Program + factor 1 (Experimental): In this "arm" one factor is set to "active" (i.e. yes):
  - diagnostic interview
  Interventions: Behavioral: HERMES (Online Self-Help Intervention based on problem-solving therapy)
- Online-Program + factors 2,3,4 (Experimental): In this "arm" three factors are set to "active" (i.e. yes):
  * motivational module
  * guidance
  * e-mail reminders
  Interventions: Behavioral: HERMES (Online Self-Help Intervention based on problem-solving therapy)
- Online-Program + factors 2,3 (Experimental): In this "arm" two factors are set to "active" (i.e. yes):
  * motivational module
  * guidance
  Interventions: Behavioral: HERMES (Online Self-Help Intervention based on problem-solving therapy)
- Online-Program + factors 2,4 (Experimental): In this "arm" two factors are set to "active" (i.e. yes):
  * motivational module
  * e-mail reminders
  Interventions: Behavioral: HERMES (Online Self-Help Intervention based on problem-solving therapy)
- Online-Program + factor 2 (Experimental): In this "arm" one factor is set to "active" (i.e. yes):
  - motivational module
  Interventions: Behavioral: HERMES (Online Self-Help Intervention based on problem-solving therapy)
- Online-Program + factors 3,4 (Experimental): In this "arm" two factors are set to "active" (i.e. yes):
  * guidance
  * e-mail reminders
  Interventions: Behavioral: HERMES (Online Self-Help Intervention based on problem-solving therapy)
- Online-Program + factor 3 (Experimental): In this "arm" one factor is set to "active" (i.e. yes):
  - guidance
  Interventions: Behavioral: HERMES (Online Self-Help Intervention based on problem-solving therapy)
- Online-Program + factor 4 (Experimental): In this "arm" one factor is set to "active" (i.e. yes):
  - e-mail reminders
  Interventions: Behavioral: HERMES (Online Self-Help Intervention based on problem-solving therapy)
- Online-Program + no factor (Experimental): In this "arm" no factor is set to "active" (i.e. yes):
  Interventions: Behavioral: HERMES (Online Self-Help Intervention based on problem-solving therapy)

INTERVENTIONS:
Behavioral: HERMES (Online Self-Help Intervention based on problem-solving therapy) — The Online Self-Help Intervention is an online program based on the problem-solving therapy (an evidence based approach of psychotherapy). All participants will receive the exact same intervention.
  However, what will be experimentally varied are the four listed interventions.
  Other Names: diagnostic telephone interview (yes/no) (prior to the access to HERMES); motivational module (yes/no) (prior to the access to HERMES); guidance (yes/no) (during the usage of HERMES); e-mail reminders (yes/no) (during the usage of HERMES)

SUMMARY:
A vast amount of studies show that online interventions are suitable to reduce symptoms of mental illness as for instance depression or anxiety. However, participants who use online interventions are more likely to drop out of treatment compared to face-to-face interventions. It is important to enhance adherence to online interventions so that participants engage longer in the programs. Also, as online interventions are useful to reduce the burden of mental illness, it is of interest to further improve outcomes of such interventions. Therefore, it will be investigated in this study whether or not four different factors have an impact in fostering adherence to and improving outcome of an internet-based self-help intervention based on problem-solving therapy. A multifactorial design will be used for this study to screen simultaneously whether or not i) a diagnostic telephone interview and, ii) an educational module based on motivational interviewing prior to the intervention and iii) guidance by the study team, and iv) automated e-mail reminders during the study are active factors in enhancing adherence to and outcome of online interventions.

ELIGIBILITY:
Inclusion Criteria:

* PHQ-9-Score between 5 - 14
* Signed Informed Consent
* Contact information provided in case of emergency
* Internet connection and device to use it (Smartphone, Computer, Tablet)
* Fluent in german language

Exclusion Criteria:

* Suicidal tendencies (SBQ-R > 7)
* a current or previous diagnose of a bipolar or psychotic disorder
* a current diagnosis of severe depression or another psychological disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Change in Depressive Symptoms | Baseline
  Assessed with Patient Health Questionnaire - Depression (PHQ-9; Kroenke, Spitzer & Williams, 2001)
Change in Depressive Symptoms | 2 weeks
  Assessed with Patient Health Questionnaire - Depression (PHQ-9; Kroenke, Spitzer & Williams, 2001)
Change in Depressive Symptoms | 4 weeks
  Assessed with Patient Health Questionnaire - Depression (PHQ-9; Kroenke, Spitzer & Williams, 2001)
Change in Depressive Symptoms | 10 weeks
  Assessed with Patient Health Questionnaire - Depression (PHQ-9; Kroenke, Spitzer & Williams, 2001)
Change in Depressive Symptoms | 16 weeks
  Assessed with Patient Health Questionnaire - Depression (PHQ-9; Kroenke, Spitzer & Williams, 2001)

SECONDARY OUTCOMES:
Adherence to Intervention (1) | through study completion, an average of 16 weeks
  Assessed with the online Program. Indicator of adherence: time spent in program
Adherence to Intervention (2) | through study completion, an average of 16 weeks
  Assessed with the online Program. Indicator of adherence: clicks
Adherence to Intervention (3) | through study completion, an average of 16 weeks
  Assessed with the online Program. Indicator of adherence: number of exercises completed
Anxiety Symptoms | Baseline, 10 weeks, 16 weeks
  Assessed with Patient Health Questionnaire - Anxiety (GAD-7; Löwe et al., 2002)
Stress Symptoms | Baseline, 10 weeks, 16 weeks
  Assessed with Patient Health Questionnaire - Stress (PHQ-Stress; Löwe et al., 2002)
Health | Baseline, 10 weeks, 16 weeks
  Assessed with Short Form Health Survey (SF-12; Gandek et al., 1998)
Suicidal Tendency | Baseline, 10 weeks, 16 weeks
  Assessed with Suicide Behaviors Questionnaire - Revised (SBQ-R; Glaesmer et al., 2017)
Social Problem Solving | Baseline, 10 weeks, 16 weeks
  Assessed with Social Problem Solving Inventory Revised (SPSI-R; D'Zurilla et al., 1999)
Satisfaction with treatment | 10 weeks
  Assessed with the german version of Client Satisfaction Questionnaire CSQ-8 (Attkisson & Zwick, 1982)
Negative Effects of Psychotherapy | 10 weeks, 16 weeks
  Assessed with "Inventory for the Assessment of Negative Effects of Psychotherapy (INEP; Ladwig, Rief, & Nestoriuc, 2014)
Usability of Intervention | 10 weeks
  Assessed with System Usability Scale (SAS; Brooke, 1996)

OTHER OUTCOMES:
Credibility and Expectancy | Baseline, 2 weeks, 4 weeks
  Assessed with Credibility/Expectancy Questionnaires (CEQ; Devilly & Borkovec, 2000)
Working Alliance | Baseline, 2 weeks, 4 weeks
  Assessed with Working Alliance Inventory - for Internet Interventions (WAI-I; Gomez Penedo et al., 2019)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Berger, Prof. Dr., Principal Investigator — University of Bern
Locations (1):
- University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available, after all planned analysis have been made by the Investigators.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data: Begin 2022 Other information: when available
Access Criteria: will be decided individually

REFERENCES:
- [Derived] Bur OT, Berger T. Participant Adherence and Contact Behavior in a Guided Internet Intervention for Depressive Symptoms: Exploratory Study. JMIR Form Res. 2024 Dec 16;8:e46860. doi: 10.2196/46860. PMID 39679951
- [Derived] Bur OT, Krieger T, Moritz S, Klein JP, Berger T. Optimizing the context of support of web-based self-help in individuals with mild to moderate depressive symptoms: A randomized full factorial trial. Behav Res Ther. 2022 May;152:104070. doi: 10.1016/j.brat.2022.104070. Epub 2022 Mar 6. PMID 35306266
- [Derived] Bur OT, Krieger T, Moritz S, Klein JP, Berger T. Optimizing the Context of Support to Improve Outcomes of Internet-Based Self-help in Individuals With Depressive Symptoms: Protocol for a Randomized Factorial Trial. JMIR Res Protoc. 2021 Feb 2;10(2):e21207. doi: 10.2196/21207. PMID 33528377
- See also: Homepage of the study — https://selfhelp.psy.unibe.ch/hermes/homepage